CLINICAL TRIAL: NCT06748417
Title: Reliability of the FITLIGHT System and Acute Effects of Cognitive Training on Dual-task Performance in Hopping and Cutting Assessments
Brief Title: FITLIGHT Reliability and Acute Training Effects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Software and hardware issues in data collection cannot be resolved.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Zachary Ripic, Principal Investigator, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20241122
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Athletic Injuries
Keywords: Reaction time; neurocognitive performance; Agility training
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acute Cognitive Training Followed by Non-stimulating Rest Group (Experimental): Participants will be in this group for approximately 11-14 days
  Interventions: Device: Acute Cognitive Training; Other: Non-stimulating Rest
- Non-stimulating rest followed by acute cognitive training Group (Experimental): Participants will be in this group for approximately 11-14 days
  Interventions: Device: Acute Cognitive Training; Other: Non-stimulating Rest

INTERVENTIONS:
Device: Acute Cognitive Training — Participants will receive the intervention in person once within in the study for 30 minutes. During the intervention, participants will receive a cognitive training session consisting of an upper extremity, lower extremity, and whole-body reaction time task. The device (5 LED) will be placed in front of participants in all tasks, and participants will be asked to deactivate lights that illuminate for a period of 30 seconds with 30 seconds of rest. For the upper and lower extremity tasks, these will be repeated on both limbs. The purpose of the tasks are to pre-train reaction time in an isolated fashion, requiring participants to use either hands or feet to deactivate the lights, as well as incorporate whole-body movement in the third task along with a decision-making (color-matching) component.
  Other Names: FITLIGHT
Other: Non-stimulating Rest — Participants will receive the intervention in person once within the study for 30 minutes. During the intervention, participants will watch, while seated, a 30-minute segment of a nature documentary. The purpose of this intervention is to ensure no additional cognitive or movement training that would improve performance on the dual-task test occurs during the intended rest period.

SUMMARY:
The purpose of this study is to assess the reliability of outcomes collected using a speed and cognitive light training system. This study will also be used to understand the effects of brain training on athletic performance using the FITLIGHT System.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a Physical Activity Readiness Questionnaire
* BMI under 30

Exclusion Criteria:

* Color-blindness
* Fractures within the past year
* Musculoskeletal injury limiting sports activity within the past 6 months
* Anterior cruciate ligament (ACL) injuries within the past 5 years
* Medical conditions that do not have physician clearance to participate in exercise
* History of concussion
* Diagnosed cognitive impairments
* Untreated attention deficit/hyperactivity disorder (ADHD) or attention deficit disorder (ADD)
* Prisoners
* Pregnant women
* Smokers

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Change in Reaction Time | Up to 5 minutes before and up to 5 minutes after intervention
  Will be measured in seconds (s)
Change in Percentage of Correct Responses in Cognitive-Motor Running T-test | Up to 5 minutes before and up to 5 minutes after intervention
  Percentage of correct responses on cognitive-motor test
Change in Completion Time | Up to 5 minutes before and up to 5 minutes after intervention
  Will be measured in seconds (s)
Change in Hop distance | Up to 10 minutes before and up to 10 minutes after intervention
  Will be measured in meters (m)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary A Ripic, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No